CLINICAL TRIAL: NCT00410397
Title: The Use of Myofascial Release in Lumbopelvic Pain
Brief Title: The Use of Manual Therapy to Treat Low-Back and Hip Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: Corey Babb/ MS4, Oklahoma State University Center for Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006028
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Low Back Pain; Pain
Keywords: Low back pain; Hip pain
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Osteopathic Manipulative Medicine
  Interventions: Procedure: Osteopathic Manipulative Medicine
- B (Placebo Comparator)
  Interventions: Procedure: Sham Manipulation

INTERVENTIONS:
Procedure: Osteopathic Manipulative Medicine — Pelvic balancing, myofascial release of the anterior pelvis.
  Arms: A
Procedure: Sham Manipulation — Neutral positional, gentle palpation
  Arms: B

SUMMARY:
Low back pain (LBP) is a common problem in the adult population with many approaches to treatment, but no clear answer. One of the causes of LBP, musculoskeletal pain, can be triggered by spasm of the deep muscles of the back and pelvis. This study, therefore, focuses on treating pelvic muscle pain as a way of lessening LBP.

DETAILED DESCRIPTION:
Osteopathic manipulative medicine (OMM) is a well-researched standard of care in the treatment of low back pain (LBP). Under the heading of OMM, many different modalities exist to decrease a patient's somatic dysfunction. Among the most commonly used are high velocity (thrusting through an immobilized joint) and muscle energy (engaging a restrictive barrier using the patient's own strength).

Although a very common complaint, there is no exact etiology for LBP. Many different theories exist, including postural disturbances, leg length discrepancies, and even genetic predispositions. A study in Spine finds that among those with chronic LBP there is a subgroup of people with reduced hip flexion, and concludes that hip motion should be considered in treatment of patients with LBP. Currently, there exists no research on the manipulation of hip flexors in the treatment of LBP. This study, therefore, will test the efficacy of OMM on the deep pelvic musculature as a way of decreasing LBP.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age-older than 18 years and younger than 65 years
* Lumbopelvic pain

Exclusion Criteria:

* Cardiovascular disease (heart-failure, myocardial infarction, hypertension)
* Diabetes
* Rheumatoid Arthritis
* Osteoarthritis
* Chronic Illness
* Pregnancy-self reported
* Neurodegenerative Disease
* Osteopenia
* Osteoporosis
* Metastatic Cancer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2006-12; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Reduction in low back pain on a 1-10 scale. | Immediately following treatment.

SECONDARY OUTCOMES:
Reduction in low back pain on a 0-10 scale. | 6-8 hours after treatment.
Reduction in low back pain on a 0-10 scale. | After four weeks of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Corey R Babb, B.A., Principal Investigator — Oklahoma State University College of Osteopathic Medicine; JoAnn G Ryan, D.O., Study Director — Oklahoma State University College of Osteopathic Medicine
Locations (1):
- Oklahoma State University College of Osteopathic Medicine, Tulsa, Oklahoma, United States

REFERENCES:
- [Background] Katz JN. Lumbar disc disorders and low-back pain: socioeconomic factors and consequences. J Bone Joint Surg Am. 2006 Apr;88 Suppl 2:21-4. doi: 10.2106/JBJS.E.01273. PMID 16595438
- [Background] Licciardone JC, Brimhall AK, King LN. Osteopathic manipulative treatment for low back pain: a systematic review and meta-analysis of randomized controlled trials. BMC Musculoskelet Disord. 2005 Aug 4;6:43. doi: 10.1186/1471-2474-6-43. PMID 16080794
- [Background] Borenstein DG. Epidemiology, etiology, diagnostic evaluation, and treatment of low back pain. Curr Opin Rheumatol. 2001 Mar;13(2):128-34. doi: 10.1097/00002281-200103000-00006. PMID 11224737
- [Background] Hestbaek L, Leboeuf-Yde C, Kyvik KO. Is comorbidity in adolescence a predictor for adult low back pain? A prospective study of a young population. BMC Musculoskelet Disord. 2006 Mar 16;7:29. doi: 10.1186/1471-2474-7-29. PMID 16539740
- [Background] Hestbaek L, Larsen K, Weidick F, Leboeuf-Yde C. Low back pain in military recruits in relation to social background and previous low back pain. A cross-sectional and prospective observational survey. BMC Musculoskelet Disord. 2005 May 26;6:25. doi: 10.1186/1471-2474-6-25. PMID 15918894
- [Background] Porter JL, Wilkinson A. Lumbar-hip flexion motion. A comparative study between asymptomatic and chronic low back pain in 18- to 36-year-old men. Spine (Phila Pa 1976). 1997 Jul 1;22(13):1508-13; discussion 1513-4. doi: 10.1097/00007632-199707010-00017. PMID 9231971